CLINICAL TRIAL: NCT01531231
Title: Typical Daily Emotions, Ischemia and Repolarization in Coronary Artery Disease
Brief Title: Typical Daily Experiences, Ischemia and Repolarization in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Richard Lane (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor-Investigator, Richard Lane, MD, PhD, University of Arizona
Organization: University of Arizona (Other)
Other Study IDs: R01HL103692-01A1 (NIH)
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Behavioral
Keywords: heart disease; unstable angina; myocardial infarction; behavioral; cardiovascular; emotions
MeSH Terms: conditions — Coronary Artery Disease; Behavior; Heart Diseases; Angina, Unstable; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- YOUNG HEALTHY NO CORONARY ARTERY DISEASE: - Whether an association between typical daily experiences and recovery time varies with age; this group will be compared to the older comparison group and to previous data collected from those subjects who participated in the Long QT Syndrome study (LQTS).
- OLDER HEALTHY NO CORONARY ARTERY DISEASE: - Determine whether daily emotion influences ischemia and repolarization differentially as a function of the severity of CAD and presence of CAD when comparing CAD patients with healthy patients
- HIGH RISK CORONARY ARTERY DISEASE (CAD): - Determine whether emotion assessed randomly throughout the day is associated with myocardial ischemia
- LOW RISK CORONARY ARTERY DISEASE (CAD): - Determine whether typical daily emotion influences ischemia and repolarization differentially as a function of the severity of CAD and presence of CAD

SUMMARY:
The purpose of this study is to examine the role of every day experiences as they relate to coronary artery disease (CAD).

DETAILED DESCRIPTION:
CAD is the most common setting in which sudden cardiac death (SCD) occurs. SCD is the leading cause of death in the U.S.

In this study we propose to test the following in patients with CAD:

* Determine whether experiences assessed randomly throughout the day are associated with changes in the blood supply to your heart muscle as measured by electrical recordings from your chest.
* Determine whether typical daily experiences are associated with changes in the recovery time portion of your heart beat cycle as measured by electrical recordings from your chest.
* Determine whether changes in the recovery time portion of your heart beat cycle associated with typical daily experiences occur exclusively with changes in the blood supply to your heart muscle.
* Determine whether typical daily experiences influences blood supply and recovery time based on the severity and presence of CAD (when comparing CAD patients to healthy subjects).

ELIGIBILITY:
KEY INCLUSION CRITERIA: LOW RISK CAD SUBJECTS, EJECTION FRACTION >35%

* Proficient in English
* At least 21 years of age or older
* Stable coronary artery disease
* Willing to participant in 3 days of Holter monitor recordings and respond to surveys on a study provided smartphone

KEY EXCLUSION CRITERIA: LOW RISK CAD SUBJECTS

- Presence of bundle branch block evident on ECG

KEY INCLUSION CRITERIA: HIGH RISK CAD Subjects, Ejection Fraction <35%

* Proficient in English
* 21 years of age or older
* Have stable coronary artery disease with a documented previous myocardial infarction
* Recent ECHO, MUGA or angiography (< 5year old) reflecting a left-ventricular ejection fraction <35%
* Single or dual chamber ICD, with a back up rate of ventricular pacing at < 45 bpm
* Willing to wear a Holter monitor for 3 days and respond to surveys on a study provided smartphone

KEY EXCLUSION CRITERIA: HIGH RISK CAD, Ejection Fraction <35%

* An implanted cardiac resynchronization pacemaker with ICD (CRT-D)
* Heart rhythm artificially continuously paced
* Presence of a bundle branch block evident on any ECG

KEY INCLUSION CRITERIA: OLDER HEALTHY COMPARISON

* Proficient in English
* 51 years of age or older
* No history and evidence of ischemic heart disease
* Normal screening ECG without evidence for rhythm abnormalities, conduction abnormalities, hypertrophy, or other pathologies
* Age matched within 5 years to CAD patients
* Negative treadmill/bicycle exercise test
* Willing to wear a Holter monitor for 3 days and respond to surveys on a study provided smartphone

KEY EXCLUSION CRITERIA: OLDER HEALTHY COMPARISON

* History of ischemic heart disease (CAD),prior myocardial infarction
* History of cardiac disease

KEY INCLUSION CRITERIA: YOUNGER HEALTHY (ENROLLMENT CLOSED)

* Proficient in English
* 21 to 50 years of age
* Normal screening ECG without evidence for rhythm abnormalities, conduction abnormalities, hypertrophy, or other pathologies
* Willing to wear a Holter monitor for 3 days and respond to surveys on a study provided smartphone

KEY EXCLUSION CRITERIA: YOUNGER HEALTHY

* History of ischemic heart disease (CAD), prior myocardial infarction
* History of cardiac diseases
* Abnormal ECG

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University of Arizona Medical Center (overhead TV monitors); Cardiology Clinics; Community Centers; Primary Care Clinics; Pima Heart; Desert Cardiology; Referrals from study participants, Craig's List
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2011-06-02 (Actual); Primary Completion 2016-03-24 (Actual); Study Completion 2016-03-29 (Actual)

PRIMARY OUTCOMES:
To obtain behavioral and cardiovascular data including 4-days collection of data as study participant engages in their daily activities. | 4 days
  To determine whether typical daily emotion is associated with myocardial ischemia and repolarization changes in patients with coronary artery disease, and then determine whether the association between repolarization changes and daily emotion is related to myocardial ischemia; whether daily emotion influences ischemia and repolarization differentially as a function of severity of coronary artery disease; whether the association between daily emotion and repolarization varies in healthy volunteers. Some of these outcomes are intertwined.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Lane, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States